CLINICAL TRIAL: NCT07099560
Title: Comparison of Preemptive Analgesic Effect of Ultrasound Guided Sacral Erector Spinae Plane Block Versus Ultrasound Guided Caudal Block in Pediatric Undergoing Hypospadias Surgery
Brief Title: Ultrasound Guided Sacral Erector Spinae Plane Block Versus Ultrasound Guided Caudal Block in Pediatric Undergoing Hypospadias Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ghada Magdy Ahmed Elfekey, Resident of Anesthesia, Surgical Intensive Care and Pain Management, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 36264MS869/3/25
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Hypospadias; Caudal Block; Erector Spinae Plane Block; Pain, Postoperative
Keywords: hypospadias; nerve block; erector spinae plane block; caudal block; pain; ultra-sound
MeSH Terms: conditions — Hypospadias; Pain, Postoperative; Pain | interventions — Anesthesia, Caudal

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel assignment. Participants are randomized 1:1 after induction of anesthesia to receive either ultrasound-guided sacral erector spinae plane block or ultrasound-guided caudal epidural block. Each participant receives one procedure only (no crossover), and both groups are followed concurrently for 24 hours with standardized perioperative care. Randomization uses a computer-generated sequence with allocation concealment via sequentially numbered, opaque, sealed envelopes. Blocks are performed by an anesthesiologist not involved in postoperative assessments; outcome assessors are blinded to group assignment. Single-center study at Tanta University Hospitals.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Sacral Erector Spinae Plane Block (sESPB) (Experimental): Participants receive bilateral ultrasound-guided sacral ESPB after induction of general anesthesia. Using a high-frequency linear probe, the needle is advanced to the sacral fascial plane near the median sacral crest; after negative aspiration, bupivacaine 0.25% at 0.5-1 mL/kg (maximum total volume 20 mL) is injected. Standardized perioperative care; rescue analgesia (pethidine 0.5 mg/kg) if FLACC ≥4.
  Interventions: Procedure: Ultrasound-guided sacral erector spinae plane block (sESPB)
- Arm B - Active Comparator: Caudal Epidural Block (Experimental): Participants receive ultrasound-guided caudal epidural block after induction of general anesthesia. Needle introduced via the sacral hiatus under ultrasound; after negative aspiration, bupivacaine 0.25% at 0.5-1 mL/kg (maximum total volume 20 mL) is injected. Standardized perioperative care; rescue pethidine if FLACC ≥4.
  Interventions: Procedure: Ultrasound-guided caudal epidural block

INTERVENTIONS:
Procedure: Ultrasound-guided sacral erector spinae plane block (sESPB) — After induction of general anesthesia, bilateral sESPB is performed under ultrasound guidance. Needle advanced to the sacral interfascial plane near the median sacral crest; after negative aspiration, bupivacaine 0.25% at 0.5-1 mL/kg (max total 20 mL) is injected. Standardized perioperative care; rescue pethidine 0.5 mg/kg if FLACC ≥4.
  Other Names: sESPB; sacral ESP block
  Arms: Arm A: Sacral Erector Spinae Plane Block (sESPB)
Procedure: Ultrasound-guided caudal epidural block — After induction of general anesthesia, caudal epidural injection via sacral hiatus under ultrasound guidance; after negative aspiration, bupivacaine 0.25% at 0.5-1 mL/kg (max total 20 mL) is injected. Standardized perioperative care; rescue pethidine if FLACC ≥4.
  Other Names: Caudal epidural block (CEB); Caudal epidural anesthesia; Caudal block
  Arms: Arm B - Active Comparator: Caudal Epidural Block

SUMMARY:
Randomized, parallel-group, assessor-blinded clinical trial at Tanta University Hospitals comparing ultrasound-guided sacral erector spinae plane block (sESPB) versus ultrasound-guided caudal epidural block for postoperative analgesia in male children (1-5 years) undergoing hypospadias repair. Seventy participants will be randomized 1:1 to receive sESPB or caudal block with 0.25% bupivacaine (0.5-1 mL/kg; maximum 20 mL) after induction of general anesthesia. The primary outcome is pain over the first 24 hours, assessed using the FLACC scale at prespecified time points. Secondary outcomes include total opioid consumption, time to first rescue analgesia, postoperative nausea and vomiting, parent/guardian satisfaction, hemodynamic trends, and predefined adverse effects (e.g., motor weakness, urinary retention, respiratory depression, hematoma, infection at injection site). Perioperative care is standardized; rescue pethidine is administered when FLACC ≥4. The trial evaluates whether sESPB provides superior or comparable analgesia with fewer adverse effects than caudal block.

DETAILED DESCRIPTION:
Randomized, parallel-group, assessor-blinded clinical trial at Tanta University Hospitals comparing ultrasound-guided sacral erector spinae plane block (sESPB) versus ultrasound-guided caudal epidural block for postoperative analgesia in male children (1-5 years) undergoing hypospadias repair. Seventy participants will be randomized 1:1 to receive sESPB or caudal block with 0.25% bupivacaine (0.5-1 mL/kg; maximum 20 mL) after induction of general anesthesia. The primary outcome is pain over the first 24 hours, assessed using the FLACC scale at prespecified time points. Secondary outcomes include total opioid consumption, time to first rescue analgesia, postoperative nausea and vomiting, parent/guardian satisfaction, hemodynamic trends, and predefined adverse effects (e.g., motor weakness, urinary retention, respiratory depression, hematoma, infection at injection site). Perioperative care is standardized; rescue pethidine is administered when FLACC ≥4. The trial evaluates whether sESPB provides superior or comparable analgesia with fewer adverse effects than caudal block.

ELIGIBILITY:
Inclusion Criteria

* Male children aged 1-5 years
* ASA physical status I-II
* Scheduled for elective hypospadias repair under general anesthesia
* Parent or legal guardian provides written informed consent
* Able to complete postoperative assessments through 24 hours after surgery Exclusion Criteria
* Parent/guardian refusal of participation
* Coagulopathy or current anticoagulant therapy
* Infection at the intended injection site (sacral/caudal region) or systemic infection
* Allergy/hypersensitivity to amide local anesthetics (e.g., bupivacaine) or study medications
* Neurologic or spinal disorders or congenital sacral anomalies affecting block safety
* Significant hepatic, renal, or cardiac disease
* Any other condition that, in the investigator's judgment, contraindicates caudal block or sacral ESPB or could interfere with safe participation

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male only. Enrollment is limited to pediatric patients with male genitalia (sex assigned male at birth) undergoing hypospadias repair. Rationale: hypospadias is a congenital condition of the penis and occurs in males; therefore, females and other genders are not eligible."
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
FLACC pain score (0-10) during the first 24 hours after surgery | From immediately after surgery through 24 hours postoperatively: at the time of Post-Anesthesia Care Unit (PACU) arrival (0 hours), and at 30 minutes, 2 hours, 4 hours, 6 hours, 12 hours, and 24 hours after surgery.
  The FLACC scale (Face, Legs, Activity, Cry, Consolability) is a validated behavioral pain measure. Each category is scored 0-2; the total score ranges 0-10 with higher scores indicating more pain. Scores will be recorded at rest by a blinded outcomes assessor at the prespecified time points. Rescue analgesia is IV pethidine 0.5 mg/kg when FLACC ≥4. The primary analysis compares groups across time (mixed-effects model) and/or as the time-weighted mean over 0-24 h.

SECONDARY OUTCOMES:
Total opioid consumption (pethidine), 0-24 h (mg/kg) | From the time of arrival to the Post-Anesthesia Care Unit (0 hours) through 24 hours after surgery.
  Cumulative dose of IV pethidine given as rescue analgesia when FLACC ≥4, from PACU arrival through 24 h post-op. Sum all doses per participant; no other opioids planned. Group summaries will be reported.
Time to first rescue analgesia requirement postoperatively | From the time of arrival to the Post-Anesthesia Care Unit (0 hours) until the first rescue dose, within 24 hours after surgery
  If FLACC pain score ≥ 4 I.V pethidine 0.5 mg/kg will be given as rescue analgesia.
Parent's satisfaction | 24 hours postoperatively
  Parent's Satisfaction Level were recorded on a numerical scale from 1 to 3 (not satisfied - neutral - satisfied).
Incidence of postoperative adverse events | 24 hours postoperatively
  Postoperative adverse events as nausea and vomiting, motor weakness, urinary retention, drowsiness, respiratory depression, hematoma or infection at the site of injection will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada MA Elfekey, MBBCH, Principal Investigator — Faculty of Medicine, Tanta University, Egypt
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia Govenorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author